CLINICAL TRIAL: NCT05831163
Title: A Review of Clinical Trial Experiences and Trends From Spinal Cord Injury Patients
Brief Title: Analyzing Clinical Research Participation of Patients With Spinal Cord Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83050803
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Spinal Cord Injuries
Keywords: Spinal Cord Injuries; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The percentages of participants in clinical studies haven't always been perfectly representative of a particular group.

This research examines the variables that affect a patient's choice to enroll in, discontinue participation in, or resume participation in a clinical trial for spinal cord injury.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future spinal cord injury research.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Ability to understand and the willingness to sign a written informed consent document.
* Diagnosis of spinal cord injury

Exclusion Criteria:

* Is pregnant, breastfeeding or expecting to conceive within the projected duration of the study
* Has a serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are actively considering involvement in an observational spinal cord injury clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a spinal cord injury clinical study. | 3 months
Number of spinal cord injury study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duan R, Qu M, Yuan Y, Lin M, Liu T, Huang W, Gao J, Zhang M, Yu X. Clinical Benefit of Rehabilitation Training in Spinal Cord Injury: A Systematic Review and Meta-Analysis. Spine (Phila Pa 1976). 2021 Mar 15;46(6):E398-E410. doi: 10.1097/BRS.0000000000003789. PMID 33620185
- [Background] Yamazaki K, Kawabori M, Seki T, Houkin K. Clinical Trials of Stem Cell Treatment for Spinal Cord Injury. Int J Mol Sci. 2020 Jun 2;21(11):3994. doi: 10.3390/ijms21113994. PMID 32498423
- [Background] Kim YH, Ha KY, Kim SI. Spinal Cord Injury and Related Clinical Trials. Clin Orthop Surg. 2017 Mar;9(1):1-9. doi: 10.4055/cios.2017.9.1.1. Epub 2017 Feb 13. PMID 28261421

DOCUMENTS (1):
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/63/NCT05831163/ICF_000.pdf